CLINICAL TRIAL: NCT06585423
Title: Tolerability of an Anesthesia-free Tonometer Tip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00115919; 399000397 (Other Grant/Funding Number: Gilhuly Accelerator Fund)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Intraocular pressure measurements using 4 different prototype tips. All standard equipment used to perform Goldmann Applanation Tonometry will be used with the only difference being the applanator tip. The 4 prototypes are as follows and are tested in random order:
  1. - Medical grade acrylic tip covered by a sterile commercially available bandage contact lens (Air Optix, Night and Day Contacts, Alcon). The bandage contact lens will be changed between subjects and the underlying acrylic tip sterilized per standard clinical procedure (bleach soak followed by soak and rinse in sterile water).
  2. - Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm. T
  3. - Medical grade acrylic tip coated with medical grade silicone of a thickness > 100 µm.
  4. - Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm with blur tint. All tips will be sterilized between subjects
  5. - Standard tip in conjunction with a topical anesthetic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Medical grade acrylic tip covered by a sterile commercially available bandage contact lens (Experimental)
  Interventions: Diagnostic Test: Sterile commercially available bandage contact lens
- Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm (Experimental)
  Interventions: Diagnostic Test: Medical grade silicone of a thickness <100 µm
- Medical grade acrylic tip coated with medical grade silicone of a thickness > 100 µm (Experimental)
  Interventions: Diagnostic Test: Medical grade silicone of a thickness >100 µm
- Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm with blue tint (Experimental)
  Interventions: Diagnostic Test: Medical grade silicone of a thickness <100 µm with blur tint
- Standard tip in conjunction with a topical anesthetic (Active Comparator)
  Interventions: Diagnostic Test: Standard tip in conjunction with a topical anesthetic

INTERVENTIONS:
Diagnostic Test: Sterile commercially available bandage contact lens — Medical grade acrylic tip covered by a sterile commercially available bandage contact lens
  Arms: Medical grade acrylic tip covered by a sterile commercially available bandage contact lens
Diagnostic Test: Medical grade silicone of a thickness <100 µm — Medical grade acrylic tip coated with medical grade silicone of a thickness <100 µm
  Arms: Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm
Diagnostic Test: Medical grade silicone of a thickness >100 µm — Medical grade acrylic tip coated with medical grade silicone of a thickness >100 µm
  Arms: Medical grade acrylic tip coated with medical grade silicone of a thickness > 100 µm
Diagnostic Test: Medical grade silicone of a thickness <100 µm with blur tint — Medical grade acrylic tip coated with medical grade silicone of a thickness <100 µm with blur tint
  Arms: Medical grade acrylic tip coated with medical grade silicone of a thickness < 100 µm with blue tint
Diagnostic Test: Standard tip in conjunction with a topical anesthetic — Standard tip in conjunction with a topical anesthetic
  Arms: Standard tip in conjunction with a topical anesthetic

SUMMARY:
The purpose of this study is to compare the tolerability and comfort of 4 different prototype anesthesia-free tonometer tips with the standard tonometer tip in conjunction with anesthesia. The best-tolerated prototype anesthesia-free tonometer tip will be identified for further development for home tonometry.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for a routine eye exam
* ≥ 18 years of age
* Able and willing to give consent

Exclusion Criteria:

* History of corneal scarring
* Active infection of the eye
* History of alternated corneal sensitivity
* History of corneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Patient tolerability rating of different tips | Baseline
  Tolerability of the different prototype anesthesia-free tonometer tips with the standard tonometer tip - based on a 0-5 scale the participants reports with higher score meaning more comfortable.
Patient comfort rating of different tips | Baseline
  Comfort of the different prototype anesthesia-free tonometer tips with the standard tonometer tip - based on a 0-5 scale the participants reports with higher score meaning more comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wen, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No